CLINICAL TRIAL: NCT03512301
Title: CAMCI: Advancing the Use of Computerized Screening in Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychology Software Tools, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amy Eschman, Grants Administration Manager, Psychology Software Tools, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13; 2SB1AG037357-04A1 (NIH)
Record Dates: First submitted 2018-04-17; First posted 2018-04-30 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Dysfunction; Cognitive Impairment; Cognitive Decline; Cognitive Change
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CAMCI Validation (Experimental): Completion of computerized tasks (Computer Assessment of Memory and Cognitive Impairment) and traditional neuropsychological tests administered via paper-pencil method by a trained administrator
  Interventions: Device: CAMCI; Diagnostic Test: MoCA; Diagnostic Test: Clinical Adjudication

INTERVENTIONS:
Device: CAMCI — CAMCI is a computerized screening tool for the assessment of cognitive status. CAMCI accurately assesses cognitive performance using standard neuropsychological tests of memory, attention, and executive ability modified for computer administration, and an innovative Virtual Environment task, testing domains such as incidental memory, not easily assessed using paper-pencil tests. Computer-administered tasks ensure standard administration and scoring, avoiding inter-site and inter-examiner variability. The CAMCI battery consists of tasks testing multiple aspects of cognitive function, and a series of self-report questions administered via tablet computer. Using touchscreen technology for response input, CAMCI takes approximately 15-20 minutes to complete.
  Other Names: Computer Assessment of Memory and Cognitive Impairment
Diagnostic Test: MoCA — The Montreal Cognitive Assessment (MoCA) is a rapid screening tool used to detect mild cognitive impairment (MCI), assessing cognitive domains (visuospatial skills, executive function, memory, attention, language, and orientation). Individual test scores are summed into a total score from 0 (worst) to 30 (best). Individuals may achieve any score within that range. Individual test scores are not reported.
  Scores:
  26-30 considered Normal; 19-25 may suggest Mild Cognitive Impairment (MCI); 10-18 can suggest moderate impairment; < 10 may indicate severe impairment
  Other Names: Montreal Cognitive Assessment
Diagnostic Test: Clinical Adjudication — Cognitive status assessed by traditional neuropsychological tests measuring visuospatial skills, executive function, memory, attention, language, orientation. Results compared to age-adjusted norms, reviewed by expert neuropsychologists for consensus classification, per Univ of Pittsburgh Alzheimers Disease Research Ctr and Ntl Alzheimers Coordinating Ctr, and Alzheimer's Assoc criteria. Final classification adjusted per clinical judgment.
  Impaired: ≥3 scores ≥2SD below norms Indeterminate: ≤2 scores >1SD below norms Normal: Neither criteria met. Total and domain scores not reported.
  Other Names: Neuropsychological Tests

SUMMARY:
Cognitive impairment is a significant health problem in the United States, resulting in costs over $100 billion a year. We will provide an efficient, effective, and financially intelligent solution to Primary Care Physician's to identify cognitive impairment in the earliest stages, delay progression through appropriate treatment, and to afford patients the opportunity to make future plans at a time when symptoms are mild and patients are able to make informed decisions concerning financial and life activities. This has the potential to delay devastating effects of cognitive impairment, and to lessen the financial burden on the health care system in the United States.

DETAILED DESCRIPTION:
Cognitive dysfunction in the elderly population, ranging from simple forgetfulness to a diagnosis of Alzheimer's disease, can impact one's quality of life and ability to function in daily activities. It is crucial that decline be detected as early as possible in order to evaluate whether the cause is treatable, and to employ appropriate treatment, if applicable. The majority of older patients rely on their primary care physician for the bulk of their healthcare needs, but there is a lack of sensitive tools available, and there is a lack of physician's time to use the tools, leading to a failure to provide therapeutic intervention at the earliest stages of loss to potentially slow the progression of disease. Psychology Software Tools, Inc. (PST) has developed the Computer Assessment of Memory and Cognitive Impairment (CAMCI), a computerized screening tool for detection of early signs of cognitive decline, which has been shown to be more effective in the identification of patients with subtle cognitive loss than the tools most frequently used within the primary care physician (PCP) office. CAMCI would provide an option for PCPs and clinicians to provide therapeutic intervention prior to a diagnosis of dementia. Recent additions to Current Procedural Terminology (CPT) codes permit insurance reimbursement for neuropsychological testing by a computer, including time for the physician's or clinical psychologist's interpretation and reporting. The introduction of this new revenue stream for PCPs and clinicians, coupled with the characteristics of being brief and self-administered make CAMCI an attractive option for improving early intervention, providing an intelligent business solution for healthcare professionals, and a useful and effective tool that allows physicians to better evaluate and serve their patients. The specific aims included in the current project focus on activities required to successfully move CAMCI to commercialization by extending support for late stage research and product development, including regulatory strategy and intellectual property development, data collection to replicate key studies, product extension through increasing minority representation, and development of a measure of meaningful change. The ultimate goal is to streamline commercialization of CAMCI, and to provide a useful and effective tool in the detection of cognitive dysfunction to physicians, the providers of the majority of healthcare to the elderly population, to improve efficiency and effectiveness of clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adequate visual and auditory acuity to allow neuropsychological testing
* Able to read, write and understand study and test requirements
* Within the age range of 60+

Exclusion Criteria:

* Significant neurologic disease, such as multi-infarct dementia, Parkinson's disease, epilepsy, stroke, multiple sclerosis or head trauma
* History of major depression or other major psychiatric disorder, such as, schizophrenia and bipolar disorder
* History of consuming 5 or more alcoholic drinks per day on a regular basis
* Montreal Cognitive Assessment (MoCA) score <10

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Zuccolotto, Study Director — Psychology Software Tools
Locations (4):
- United States (4):
  - Indiana University, Indianapolis, Indiana
  - Psychology Software Tools, Sharpsburg, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Quality-controlled raw data as well as processed data used in publications will be made available. Shared data will include computerized task scores, neuropsychological test scores, and full analytical codes used to process and analyze the data. Workflows will be described and documented to allow replication of results from the raw data.
  Data and corresponding documentation will be made available through Open Science Framework, in addition to any potential requirements on software sharing by journals.
  The PI or Co-Investigators will disseminate results from this research through presentations at public lectures, scientific institutions and meetings, and/or publication in major journals. The PI and Co-Investigators will adhere to the NIH Grants Policy on Sharing of Unique Research Resources including the Sharing of Biomedical Research Resources: Guidelines for Recipients of NIH Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be deposited into the repository indicated above as soon as possible, but no later than 4 years after the end of the award project period.
  The Small Business Act provides authority for NIH to protect from disclosure and nongovernmental use all Small Business Innovative Research (SBIR) data developed from work performed under an SBIR funding agreement for a period of 4 years after the closeout of either a phase I or phase II grant unless NIH obtains permission from the awardee to disclose these data. The data rights protection period lapses only upon expiration of the protection period applicable to the SBIR award, or by agreement between the small business concern and NIH.
Access Criteria: PST will identify where the data will be available and how to access the data in any publications and presentations about these data, as well as acknowledge the repository and funding source in any publications and presentations. In addition, PST will abide by the policies and procedures required by the repository indicated above, fully consistent with NIH data sharing policies and applicable laws and regulations.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Recruitment occurred at 4 participating sites representing a variety of regions across the US
  * Participants were recruited from both clinical and community settings.
  * Participants were required to be at least 60 years of age, have adequate visual and auditory acuity to allow neuropsychological tests
  * Exclusionary criteria included significant neurologic disease, history of major depression, psychiatric disorder, consuming 5 or more alcoholic drinks per day, MoCA score less than 10
Groups:
- CAMCI Validation: Validation of the Computer Assessment of Memory and Cognitive Impairment (CAMCI) against 1) clinical adjudication of traditional neuropsychological tests administered via paper and pencil and 2) the Montreal Cognitive Assessment (MoCA) tool for early detection of mild cognitive impairment (MCI)
Period: Overall Study
Arm/Group | CAMCI Validation
Started | 773
Completed | 764
Not Completed | 9
Not completed — Protocol Violation | 2
Not completed — Did Not Qualify | 3
Not completed — Age-ineligible | 1
Not completed — Inadequate fluency with the English language | 3

BASELINE CHARACTERISTICS:
Arm/Group | CAMCI Validation
Number analyzed (Participants) | 764
Age, Continuous [Mean (Full Range); unit: years] — 60 years or older
  years | 71.0 [60 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 550
  Male | 214
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 116
  Not Hispanic or Latino | 619
  Unknown or Not Reported | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 266
  White | 434
  More than one race | 43
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 764
Neuropsychological classification [Count of Participants; unit: Participants] — Cognitive status assessed by traditional neuropsychological tests measuring visuospatial skills, executive function, memory, attention, language, orientation. Results compared to age-adjusted norms, reviewed by expert neuropsychologists for consensus classification, per Univ of Pittsburgh Alzheimers Disease Research Ctr and Ntl Alzheimers Coordinating Ctr, and Alzheimer's Assoc criteria. Final classification adjusted per clinical judgment.
  Impaired: ≥3 scores ≥2SD below norms Indeterminate: ≤2 scores >1SD below norms Normal: Neither criteria met. Total and domain scores not reported.
  Participants
    Normal | 521
    Indeterminate | 176
    Impaired | 67
Montreal Cognitive Assessment (MoCA) [Count of Participants; unit: Participants] — The Montreal Cognitive Assessment (MoCA) is a rapid screening tool to detect mild cognitive impairment (MCI), assessing cognitive domains (visuospatial skills, executive function, memory, attention, language, and orientation). Individual subtest scores are summed for a total score from 0 (worst) to 30 (best). Individuals may achieve any score within that range. Individual subtest scores are not reported.
  Score range with Classification: 26-30 considered Normal; 19-25 may suggest Mild Cognitive Impairment (MCI); 10-18 can suggest moderate impairment; < 10 may indicate severe impairment
  Participants
    Normal (Score Range 26-30) | 337
    Indeterminate (Score Range 19-25) | 388
    Impaired (Score Range 10-18) | 39
CAMCI [Count of Participants; unit: Participants] — CAMCI (Computer Assessment of Memory and Cognitive Impairment) is a screening tool for assessment of cognitive status using neuropsychological tests of memory, attention, executive ability modified for computer administration, and a Virtual Environment task assessing cognitive areas not easily assessed by paper tests. Score is a weighted sum of individual task scores converted to total score from 0-worst to 50-best. Intended use provides single score/cognitive classification. Individual task scores not reported. Score Range with Classification: 21-50=Normal, 16-20=Indeterminate, 0-15=Impaired
  Participants
    Normal (Score Range 21-50) | 596
    Indeterminate (Score Range 16-20) | 96
    Impaired (Score Range 0-15) | 72
WRAT5 - Word Reading [Mean (Standard Deviation); unit: points] — The Wide Range Achievement Test, 5th Edition (WRAT5), Word Reading test assess fundamental reading skills and can indicate cognitive impairments affecting academic performance. Participant reads aloud a list of letters (15) and words (55). One point for each letter or word read correctly. Higher scores are better. Score range 0-70 points.
  points | 59.59 (8.33)
WAIS-IV Digit Span Forward [Mean (Standard Deviation); unit: points] — The Digit Span Forward (DSF) (Wechsler et al., 1987), part of the Wechsler Adult Intelligence Scale, 4th Edition (WAIS-IV) evaluates short-term memory and attention. Examiner reads a span of digits at a rate of one digit per second. Participant must repeat the digits back to the examiner in sequential (forward) order. Two trials are presented at each span length. The length of span is increased (Max Span 0-9) if at least 1 correct response given at the current span length. A point is awarded for each correct recall. Score is the total points obtained (0-16). Higher scores are better.
  points
    Max Span (0-9) - number of digits recalled on the final correct trial | 6.23 (1.30)
    Score (0-16) - total of points obtained on each trial/span (0,1,2) | 9.42 (2.23)
WAIS-IV Digit Span Backward [Mean (Standard Deviation); unit: points] — The Digit Span Backward (DSB) (Wechsler et al., 1987), part of the Wechsler Adult Intelligence Scale, 4th Edition (WAIS-IV) evaluates working memory and cognitive flexibility. Examiner reads a span of digits at a rate of one digit per second. Participant must repeat the digits back to the examiner in reverse (backward) order. Two trials are presented at each span length. The length of span is increased (Max Span 0-8) if at least 1 correct response given at the current span length. A point is awarded for each correct recall. Score is the total points obtained (0-16). Higher scores are better.
  points
    Max Span (0-8) - number of digits recalled on the final correct trial | 4.40 (1.34)
    Score (0-16) - total of points obtained on each trial/span (0,1,2) | 7.77 (2.36)
WMS-IV Logical Memory I - Immediate Recall [Mean (Standard Deviation); unit: points] — The Logical Memory I, part of the Wechsler Memory Scale, 4th Edition (WMS-IV), Wechsler (1987), evaluates immediate verbal memory recall and the ability to encode and retrieve information quickly. Participant is read 2 short stories selected by age (Adult=60-69 years old, Older Adult=65-90 years old) and asked to recall as many details as possible immediately after hearing each story. Score is the number of details correctly recalled (1 point per correct detail.) Scores range based on story complexity (0-14, or 0-25). Story scores are summed for a Total Score. Population: The standardized test is provided in two forms that are selected based on participant age and ability. The age groups for this study are adults ages 60 to 69 years old and older adults ages 65 to 90 years old. There were 355 participants assigned to the adult group and 409 participants assigned to the older adult group.
  points
    Story A 1st Immediate Recall (older adult), Score Range (0-14): number analyzed (Participants) | 409
    Story A 1st Immediate Recall (older adult), Score Range (0-14) | 8.59 (2.72)
    Story A 2nd Immediate Recall (older adult), Score Range (0-14): number analyzed (Participants) | 409
    Story A 2nd Immediate Recall (older adult), Score Range (0-14) | 11.16 (2.94)
    Story B Immediate Recall (older adult), Score Range (0-25): number analyzed (Participants) | 409
    Story B Immediate Recall (older adult), Score Range (0-25) | 11.52 (4.68)
    Immediate Recall Total (older adult), Score Range (0-53): number analyzed (Participants) | 409
    Immediate Recall Total (older adult), Score Range (0-53) | 31.27 (8.69)
    Story B Immediate Recall (adult), Score Range (0-25): number analyzed (Participants) | 355
    Story B Immediate Recall (adult), Score Range (0-25) | 13.48 (4.17)
    Story C Immediate Recall (adult), Score Range (0-25): number analyzed (Participants) | 355
    Story C Immediate Recall (adult), Score Range (0-25) | 11.84 (3.86)
    Immediate Recall Total (adult), Score Range (0-50): number analyzed (Participants) | 355
    Immediate Recall Total (adult), Score Range (0-50) | 25.32 (7.36)
WMS-IV Logical Memory II - Delayed Recall [Mean (Standard Deviation); unit: points] — The Logical Memory II, part of the Wechsler Memory Scale, 4th Edition (WMS-IV), Wechsler (1987), evaluates delayed memory recall, which involves the ability to store information and retrieve it after a period of time. Participant is read 2 short stories selected by age (Adult=60-69 years old, Older Adult=65-90 years old). After a delay of ~30 minutes, participant is asked to recall as many details as possible. Score is the number of details correctly recalled (1 point per correct detail.) Scores range based on story complexity (0-14, or 0-25). Story scores are summed for a Total Score. Population: The standardized test is provided in two forms that are selected based on participant age and ability. The age groups for this study are adults ages 60 to 69 years old and older adults ages 65 to 90 years old. There were 355 participants assigned to the adult group and 409 participants assigned to the older adult group.
  points
    Story A Delayed Recall (older adult), Score Range (0-14): number analyzed (Participants) | 409
    Story A Delayed Recall (older adult), Score Range (0-14) | 7.94 (3.72)
    Story B Delayed Recall (older adult), Score Range (0-25): number analyzed (Participants) | 409
    Story B Delayed Recall (older adult), Score Range (0-25) | 9.99 (5.09)
    Delayed Recall Total (older adult), Score Range (0-39): number analyzed (Participants) | 409
    Delayed Recall Total (older adult), Score Range (0-39) | 17.93 (8.10)
    Story B Delayed Recall (adult), Score Range (0-25): number analyzed (Participants) | 355
    Story B Delayed Recall (adult), Score Range (0-25) | 11.57 (4.69)
    Story C Delayed Recall (adult), Score Range (0-25): number analyzed (Participants) | 355
    Story C Delayed Recall (adult), Score Range (0-25) | 10.37 (4.28)
    Delayed Recall Total (adult), Score Range (0-50): number analyzed (Participants) | 355
    Delayed Recall Total (adult), Score Range (0-50) | 21.93 (8.27)
Rey-Osterrieth Complex Figure Test (ROCF) [Mean (Standard Deviation); unit: points] — The Rey-Osterrieth Complex Figure Test (ROCF) (Meyers and Meyers, 1995), evaluates visuospatial abilities, memory, attention, and executive functions. Participant is presented with a complex geometric figure to study then reproduce the figure on a blank sheet of paper. After ~3 minutes (immediate recall) and ~30 minutes (delayed recall) participant must reproduce the figure again from memory. Each reproduction is scored based on 18 design elements with 0, .5, 1, or 2 points awarded per element based on element accuracy and placement.
  points
    Figure Copy | 28.31 (5.61)
    Immediate Recall - Short Delay (3 minutes) | 13.24 (5.99)
    Delayed Recall - Long Delay (30 minutes) | 12.99 (5.98)
Letter Fluency (F-A-S) Test [Mean (Standard Deviation); unit: points] — The Letter Fluency (F-A-S) Test, a subtest of the Neurosensory Center Comprehensive Examination for Aphasia (Spreen and Benton, 1977) evaluates phonemic verbal fluency and can assess language abilities, executive functions, and cognitive flexibility. Participant is asked to generate as many words as possible that begin with the letters "F," "A," and "S" within 60 seconds for each letter. Score is total words generated (1 point per unique word) within the time limit. Higher scores are better. There is no fixed upper limit of the score.
  points
    Fluency - F | 12.52 (4.49)
    Fluency - A | 11.17 (4.67)
    Fluency - S | 13.61 (4.92)
    Fluency Total | 37.29 (12.70)
Semantic Fluency Test (Animals) [Mean (Standard Deviation); unit: points] — The Semantic Fluency Test (animals) (Spreen and Strauss, 1997), evaluates semantic memory, language abilities, and executive functions, including cognitive flexibility and retrieval from long-term memory. Participant is asked to name as many animals as they can within 60 seconds. Score is total animal names generated (1 point per unique animal named) within the time limit. Higher scores are better. There is no fixed upper limit of the score.
  points | 18.65 (5.15)
Hopkins Verbal Learning Test - Revised (HVLT-R) - Recall [Mean (Standard Deviation); unit: points] — The Hopkins Verbal Learning Test - Revised (HVLT-R) evaluates verbal learning and memory. Participant is presented with a list of 12 nouns, 4 words each from 3 semantic categories and asked to recall them over a series of 3 Learning Trials. Score ranges 0-12 on each trial (1 point per each correct word). The score from each trial is summed for a Learning Trials Total Recall Score (0-36). After a 20 minute delay, the participant performs a final recall for a Delayed Recall Score (0-12). Higher is better for all scores. Retention % = Delayed Recall score / high score from Learning Trials 2 or 3.
  points
    Learning Trial 1 Recall | 5.46 (1.85)
    Learning Trial 2 Recall | 7.68 (2.16)
    Learning Trial 3 Recall | 8.82 (2.28)
    Learning Trials Total Recall | 21.96 (5.70)
    Delayed Recall (20 minutes) | 7.25 (3.21)
Hopkins Verbal Learning Test - Revised (HVLT-R) - Retention % [Mean (Standard Deviation); unit: percentage] — The Hopkins Verbal Learning Test - Revised (HVLT-R) evaluates verbal learning and memory. Participant is presented 12 nouns, 4 words each from 3 semantic categories and asked to recall them over a series of 3 Learning Trials. Score ranges 0-12 on each trial (1 point per correct word). The score from each trial is summed for a Learning Trials Total Recall Score (0-36). After a 20 minute delay, participant performs a final recall for a Delayed Recall Score (0-12). Retention % = Delayed Recall score / high score from Learning Trials 2 or 3. Higher Retention % is better, as is not capped to 100%.
  percentage | 77.77 (28.47)
Trail Making Test - Score [Mean (Standard Deviation); unit: points] — The Trail Making Test (TMT) (Reitan et al., 1958) evaluates processing speed, attention, and executive function. Participant draws lines as instructed to connect 25 circles labeled with numbers or letters without lifting the pen. One point awarded per correct line drawn (0-24, higher is better.) Task completion time is recorded in seconds. In Part A participant has 150 seconds to connect the numbered circles in ascending order (1-2-3, etc.). In Part B participant has 300 seconds to connect 25 circles alternating between numbers and letters in ascending order (1-A-2-B, etc.)
  points
    Part A Score | 24.00 (0.05)
    Part B Score | 23.54 (2.45)
Hopkins Verbal Learning Test - Revised (HVLT-R) - Recognition [Mean (Standard Deviation); unit: count] — The Hopkins Verbal Learning Test - Revised (HVLT-R) evaluates verbal learning and memory. Participant is presented 12 nouns and asked to recall them over 3 Learning Trials followed by a 20 minute Delayed Recall. Participant is then presented 12 target + 12 distractor words (6 semantically related, 6 semantically unrelated) and asked to recognize any prior words presented. Retention % = Delayed Recall score divided by high score from Learning Trials 2 or 3. Retention Discrimination Index (-12 to 12) is calculated as number of true-positives - number of false positives. Higher scores are better.
  count
    Recognition - True Positives | 10.94 (1.45)
    Recognition - False Positives | 1.42 (1.61)
    Recognition Discrimination Index | 9.53 (2.30)
Trail Making Test - Completion Time [Mean (Standard Deviation); unit: time in seconds] — The Trail Making Test (TMT) (Reitan et al., 1958) evaluates processing speed, attention, and executive function. Participant draws lines as instructed to connect 25 circles labeled with numbers or letters without lifting the pen. One point awarded per correct line drawn (0-24, higher is better.) Task completion time is recorded in seconds. In Part A participant has 150 seconds to connect the numbered circles in ascending order (1-2-3, etc.). In Part B participant has 300 seconds to connect 25 circles alternating between numbers and letters in ascending order (1-A-2-B, etc.)
  time in seconds
    Part A Time (150 seconds max) | 37.28 (18.79)
    Part B Time (300 seconds max) | 106.16 (63.65)
WAIS-IV Digit Symbol Substitution Test (DSST) [Mean (Standard Deviation); unit: points] — The Digit Symbol Substitution Test (DSST) part of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) (Wechsler et al., 1987) evaluates processing speed, attention, and motor skills. Performance correlates with real-world functional outcomes e.g., ability to accomplish everyday tasks. Participant is given a sheet of numbers and a key showing a unique symbol corresponding to each number. Participants match symbols to numbers by copying the correct symbol into spaces below each number within 120 seconds. Higher scores are better. Score range 0-135, 1 point for each correct symbol matched.
  points | 52.36 (15.45)
Boston Naming Test [Mean (Standard Deviation); unit: points] — The Boston Naming Test (BNT) 2nd edition (Kaplan et al., 2000) evaluates language abilities, specifically confrontation naming. Participant is shown 60 black-and-white line drawings of objects, one at a time for up to 20 seconds and asked to name each object. If participant struggles to name an object, examiner can provide a stimulus cue (descriptive) and a phonemic cue (sound-based). Score is the number of correct responses, including those given after a stimulus cue but excluding those given after a phonemic cue. Scores range from 0-60. Higher scores are better.
  points | 52.20 (7.36)

OUTCOME MEASURES:

1. Primary Outcome: Agreement Analysis (Agreement to Reference Standard) - Test Group
Description: Comparison (positive and negative percent agreement, confidence interval estimates, and quadratic weighted kappa) between CAMCI and clinical adjudication classifications for the Test group. Power calculations for agreement were assessed for Cohen Kappa's assuming at least 75% Normals with 80% power and .05 significance level, finding that we were sufficiently powered with at least 120 individuals in the test set, for a Kappa of at least 0.3.
Time Frame: baseline
Population: Test group. Of 773 participants enrolled, 9 were excluded, leaving 764 for analysis. Participants who completed CAMCI version A at baseline (N=680) were assigned through stratified random sampling to Training (75%) or Test (25%) groups, balanced by age, education, race, ethnicity, gender, and cognitive classification. The groups were further adjusted to match the racial and ethnic distribution in the U.S., resulting in a Training group (N=374) and a Test group (N=126).
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Adjudication - Normal: Participants classified as Normal through clinical adjudication.
- Clinical Adjudication - Indeterminate: Participants classified as Indeterminate through clinical adjudication.
- Clinical Adjudication - Impaired: Participants classified as Impaired through clinical adjudication.
Arm/Group | Clinical Adjudication - Normal | Clinical Adjudication - Indeterminate | Clinical Adjudication - Impaired
Number analyzed (Participants) | 87 | 33 | 6
Participants
  CAMCI - Normal (Scores 21-50) | 76 | 18 | 2
  CAMCI - Indeterminate (Sores 16-20) | 8 | 4 | 1
  CAMCI - Impaired (Scores 0-15) | 3 | 11 | 3
Statistical Analysis 1: Comparison: Clinical Adjudication - Normal vs Clinical Adjudication - Indeterminate vs Clinical Adjudication - Impaired; Test type: Other; Accuracy = 0.6587, 95% CI 2-sided [0.5690 to 0.7408]
Statistical Analysis 2: Comparison: Clinical Adjudication - Normal; Test type: Other; Sensitivity = 0.8736
Statistical Analysis 3: Comparison: Clinical Adjudication - Normal; Test type: Other; Specificity = 0.4872
Statistical Analysis 4: Comparison: Clinical Adjudication - Normal; Test type: Other; Positive Predictive Value = 0.7917
Statistical Analysis 5: Comparison: Clinical Adjudication - Normal; Test type: Other; Negative Predictive Value = 0.6333
Statistical Analysis 6: Comparison: Clinical Adjudication - Indeterminate; Test type: Other; Sensitivity = 0.1212
Statistical Analysis 7: Comparison: Clinical Adjudication - Indeterminate; Test type: Other; Specificity = 0.9032
Statistical Analysis 8: Comparison: Clinical Adjudication - Indeterminate; Test type: Other; Positive Predictive Value = 0.3077
Statistical Analysis 9: Comparison: Clinical Adjudication - Indeterminate; Test type: Other; Negative Predictive Value = 0.7434
Statistical Analysis 10: Comparison: Clinical Adjudication - Impaired; Test type: Other; Sensitivity = 0.5000
Statistical Analysis 11: Comparison: Clinical Adjudication - Impaired; Test type: Other; Specificity = 0.8833
Statistical Analysis 12: Comparison: Clinical Adjudication - Impaired; Test type: Other; Positive Predictive Value = 0.1765
Statistical Analysis 13: Comparison: Clinical Adjudication - Impaired; Test type: Other; Negative Predictive Value = 0.9725
Statistical Analysis 14: Comparison: Clinical Adjudication - Normal vs Clinical Adjudication - Indeterminate vs Clinical Adjudication - Impaired; Test type: Other; Quadratic Weighted Kappa = 0.4446, 95% CI 2-sided [0.2791 to 0.6101]

2. Primary Outcome: Agreement Analysis (Agreement to Non-Reference Standard) - Test Group
Description: Linear regression agreement analysis (linear regression equation and confidence intervals, and Pearson correlation) between CAMCI and Montreal Cognitive Assessment (MoCA) for the Test group. Comparison (positive and negative percent agreement, confidence interval estimates, and quadratic weighted kappa) between CAMCI and Montreal Cognitive Assessment (MoCA) for the Test group.
  CAMCI Scores ranged from 0-50, higher scores mean better outcome. MoCA scores ranged from 0-30, higher scores mean better outcome.
  Power calculations for agreement were assessed for Cohen Kappa's assuming at least 75% Normals with 80% power and .05 significance level, finding that we were sufficiently powered with at least 120 individuals in the test set, for a Kappa of at least 0.3.
Time Frame: baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- MoCA - Normal (Scores 26-30): Participants classified as Normal by MoCA score ranges
- MoCA - Indeterminate (Scores 19-25): Participants classified as Indeterminate by MoCA score ranges
- MoCA - Impaired (Scores 0-18): Participants classified as Impaired by MoCA score ranges
Arm/Group | MoCA - Normal (Scores 26-30) | MoCA - Indeterminate (Scores 19-25) | MoCA - Impaired (Scores 0-18)
Number analyzed (Participants) | 57 | 63 | 6
Participants
  CAMCI - Normal | 54 | 40 | 2
  CAMCI - Indeterminate | 1 | 12 | 0
  CAMCI - Impaired | 2 | 11 | 4
Statistical Analysis 1: Comparison: MoCA - Normal (Scores 26-30) vs MoCA - Indeterminate (Scores 19-25) vs MoCA - Impaired (Scores 0-18); Test type: Other — Linear Regression. Power calculations for linear regression between CAMCI and MoCA were found to be sufficiently powered with a Pearson's R of at least 0.3 at 80% power and that equated to a test-set size of 98; Pearson Correlation = 0.5073, 95% CI 2-sided [0.3892 to 0.6091] — Linear Regression Equation: [CAMCI Score] = -5.42 + 1.40 X [MoCA Score]
Statistical Analysis 2: Comparison: MoCA - Normal (Scores 26-30) vs MoCA - Indeterminate (Scores 19-25) vs MoCA - Impaired (Scores 0-18); Test type: Other; Accuracy = 0.5556, 95% CI 2-sided [0.4644 to 0.6440]
Statistical Analysis 3: Comparison: MoCA - Normal (Scores 26-30); Test type: Other; Sensitivity = 0.9747
Statistical Analysis 4: Comparison: MoCA - Normal (Scores 26-30); Test type: Other; Specificity = 0.3913
Statistical Analysis 5: Comparison: MoCA - Normal (Scores 26-30); Test type: Other; Positive Predictive Value = 0.5625
Statistical Analysis 6: Comparison: MoCA - Normal (Scores 26-30); Test type: Other; Negative Predictive Value = 0.9000
Statistical Analysis 7: Comparison: MoCA - Indeterminate (Scores 19-25); Test type: Other; Sensitivity = 0.1905
Statistical Analysis 8: Comparison: MoCA - Indeterminate (Scores 19-25); Test type: Other; Specificity = 0.9841
Statistical Analysis 9: Comparison: MoCA - Indeterminate (Scores 19-25); Test type: Other; Positive Predictive Value = 0.9231
Statistical Analysis 10: Comparison: MoCA - Indeterminate (Scores 19-25); Test type: Other; Negative Predictive Value = 0.5487
Statistical Analysis 11: Comparison: MoCA - Impaired (Scores 0-18); Test type: Other; Sensitivity = 0.6667
Statistical Analysis 12: Comparison: MoCA - Impaired (Scores 0-18); Test type: Other; Specificity = 0.8917
Statistical Analysis 13: Comparison: MoCA - Impaired (Scores 0-18); Test type: Other; Positive Predictive Value = 0.2353
Statistical Analysis 14: Comparison: MoCA - Impaired (Scores 0-18); Test type: Other; Negative Predictive Value = 0.9817
Statistical Analysis 15: Comparison: MoCA - Normal (Scores 26-30) vs MoCA - Indeterminate (Scores 19-25) vs MoCA - Impaired (Scores 0-18); Test type: Other; Quadratic Weighted Kappa = 0.3931, 95% CI 2-sided [0.2401 to 0.5461]

3. Other Pre Specified Outcome: Change Metric (Measure of Significant Change)
Description: To derive a measure of reliable change that addressed unbalanced repeated measures and unequal timing of repeat measures, we built a two-stage hierarchical model for longitudinal data using Bayesian methods. Additionally, the standard deviation (SD) was allowed to change over time, which allowed for computation of an intraclass correlation coefficient (ICC), a measure of reliability. With an SD and ICC that can change over time, reliable change was computed for follow-up months from 3 to 24, in groups of 3. Reliable change was then adjusted for practice effects according to Duff, K. (2012).
  Computer Assessment of Memory and Cognitive Impairment (CAMCI) scores were calculated as the weighted sum of individual task scores converted to a total score from 0-worst to 50-best. As the intended use of CAMCI is to provide a single score of overall cognitive status, individual task scores were not reported.
Time Frame: baseline, 6 months, 12 months, 24 months post baseline
Population: Individuals who received a consistent version of CAMCI across all visits (i.e., CAMCI-A), and were classified as Normal through clinical adjudication at all visits.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- CAMCI Baseline and Follow-Ups: Computerized and paper-pencil neuropsychological tests, baseline and CAMCI: CAMCI battery of computerized tasks
Arm/Group | CAMCI Baseline and Follow-Ups
Number analyzed (Participants) | 137
score on a scale
  0-6 Months | 11.33 [9.81 to 13.10]
  0-12 Months | 11.32 [9.79 to 13.10]
  6-24 Months | 11.38 [9.95 to 13.12]
  12-24 Months | 11.42 [10.00 to 13.18]

ADVERSE EVENTS:
Time Frame: 24 months Participants were seen at baseline only, at baseline-6 months-12 months, or at baseline-12 months-24 months. Adverse events were collected from the time a participant was enrolled until scheduled sessions were completed according to the participant's assigned group (max 24 months). COVID interruptions and project extensions, the study lasted 4 years, 4 months. Adverse events were reviewed by the Data Safety Monitoring Board as appropriate during the entire study period.
Groups:
- CAMCI Validation: Computerized and paper-pencil neuropsychological tests, baseline
  CAMCI: CAMCI battery of computerized tasks
Arm/Group | CAMCI Validation
All-Cause Mortality (participants affected / at risk) | 5/773
Serious Adverse Events (participants affected / at risk) | 6/773
Other Adverse Events (participants affected / at risk) | 1/773
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAMCI Validation (N=773)
Death unrelated to intervention reported by caregiver or test site (General disorders) | 5
Withdrawal due to health problems unrelated to intervention (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAMCI Validation (N=773)
Strain (General disorders) | 1 — One participant reported feeling tired and "strained" after completing the assessment but recovered without treatment.

LIMITATIONS AND CAVEATS:
Baseline and Follow-Up assessment targets were not reached due to suspension of the trial during the COVID-19 pandemic. Sites prohibited in-person testing for a period of 6 months, resulting in withdrawal of subjects and loss of follow-up data according to the planned timeline. Additionally, after restart, the year 3 award restricted activities during the last 6 months of the project to analysis only, limiting testing duration. By design, the trial required 36 months to complete all follow-ups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT03512301/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT03512301/SAP_001.pdf